CLINICAL TRIAL: NCT07301164
Title: A Study of BCT301 (Anti-CD19 Chemically Induced Pluripotent Stem Cell (CiPSC)-Derived CAR-iT Cells) Therapy for Refractory Autoimmune Diseases
Brief Title: Clinical Study of BCT301 Cell Injection Therapy for Refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCT301
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: System Lupus Erythematosus; Systemic Sclerosis (SSc); Inflammatory Myositis; Antiphospholipid Syndrome; ANCA Associated Vasculitis; Sjogren Syndrome
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Antiphospholipid Syndrome; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Sjogren's Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCT301 (Experimental)
  Interventions: Biological: BCT301

INTERVENTIONS:
Biological: BCT301 — BCT301, an anti-CD19 Chemically induced pluripotent stem cell (CiPSC)-derived CAR-iT cells.Participants will receive a single infusion of BCT301 cell injection at escalating dose levels.Prior to infusion, patients undergo a lymphodepleting conditioning regimen with fludarabine and cyclophosphamide given intravenously for three consecutive days.

SUMMARY:
This study primarily involves the use of BCT301, an anti-CD19 Chemically induced pluripotent stem cell (CiPSC)-derived CAR-iT cells, for the treatment of patients with refractory autoimmune diseases, aiming to evaluate its safety, tolerability, and dose-limiting toxicities(DLT), and to determine the recommended therapeutic dose for further investigation. Additionally, the study assesses the efficacy of BCT301 cell injection in refractory autoimmune diseases, as well as the pharmacokinetic (PK) and pharmacodynamic (PD) characteristics in study participants.

DETAILED DESCRIPTION:
Autoimmune diseases are a class of disorders caused by abnormal immune responses against the body's own tissues or organs. Although significant therapeutic advances have been made, such as the use of biologics (e.g., rituximab), most available drugs can only alleviate symptoms or slow disease progression, rather than achieve a complete cure.BCT301 cell injection is a CD19-targeted CAR-iT (chemically induced T-cell) therapy derived from human chemically induced pluripotent stem cells (CiPSCs) through chemical reprogramming technology. Starting from healthy donor cells, human CiPSCs are generated via small molecule-based reprogramming, followed by induced hematopoietic differentiation, iT-cell differentiation and expansion, and finally CAR lentiviral transduction to produce the off-the-shelf, CD19-targeted CAR-iT cell product (BCT301 cell injection). This approach holds promise as a potentially effective treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Voluntarily sign the informed consent form.
2. Male or female, aged 18-80 years (inclusive), with a body weight ≥40 kg.
3. Female participants of childbearing potential and male participants with female partners of childbearing potential must use medically approved contraceptive methods or practice abstinence during the treatment period and for at least 6 months after the end of the treatment. Female participants of childbearing potential must have a negative serum human chorionic gonadotropin (HCG) test within 7 days prior to enrollment and must not be breastfeeding.
4. Participants currently receiving one or more of the following treatments at stable doses: glucocorticoids, antimalarials, immunosuppressants:

   1. If the participant is receiving glucocorticoid therapy, the following conditions must be met: the maximum dose at screening and during the screening period is 30 mg/day of prednisone (or equivalent). The dose must have been stable for ≥7 days prior to screening, and adjustments during the screening period must not exceed 5 mg/day of prednisone (or equivalent);
   2. If the participant is receiving antimalarials and/or conventional immunosuppressants: the treatment must have been initiated ≥12 weeks prior to screening. The dose must have been stable for ≥8 weeks prior to screening and remain stable during the screening period;
   3. If biological agents (belimumab, telitacicept, rituximab, etc.) were used prior to the screening period, a washout period of at least 5 half-lives must be completed before screening.
5. Peripheral blood B cells must show positive CD19 expression as detected by flow cytometry.

Disease-Specific Inclusion Criteria

1. Systemic Lupus Erythematosus (SLE)

1. Meet the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE.
2. Have moderate to severe disease activity at screening, with a Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2000) score >6.
3. Have inadequate response to conventional therapy or experience disease relapse after remission. Conventional therapy includes glucocorticoids (at full or pulse doses), two or more immunosuppressants, or biologic agents for at least 6 months, including cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, leflunomide, methotrexate, belimumab, telitacicept, and rituximab.
4. Have positive serological autoantibody tests: positive antinuclear antibodies (ANAs) and/or anti-ds-DNA antibodies and/or anti-Sm antibodies.

2. Systemic Sclerosis (SSc)

1. Meet the 2013 EULAR/ACR classification criteria for SSc.
2. Fulfill either (a) or (b) below:

   1. Inadequate response to conventional therapy or disease relapse after remission. Conventional therapy includes glucocorticoids (at full or pulse doses), two or more immunosuppressants, or biologic agents for at least 6 months, including cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, leflunomide, methotrexate, belimumab, telitacicept, and rituximab.
   2. Disease progression: skin progression with a modified Rodnan Skin Score (mRSS) ≥10; and/or interstitial lung disease evidenced by ground-glass opacities on high-resolution computed tomography (HRCT); a decline in forced vital capacity (FVC) ≥10%, or a decline in FVC ≥5% accompanied by a decline in diffusing capacity for carbon monoxide (DLCO) ≥15%.
3. Have positive SSc-related autoantibodies. 3. Antiphospholipid Syndrome (APS)

1) Meet the 2006 Sydney criteria for primary antiphospholipid syndrome. 2) Have medium to high titers of antiphospholipid antibodies (lupus anticoagulant [LA], anti-β2-glycoprotein 1 [β2GP1] IgG/IgM, or anti-cardiolipin [aCL] IgG/IgM); 3) Fulfill either (a) or (b) below:

1. Receiving standard treatment with warfarin or alternative vitamin K antagonists (maintaining target international normalized ratio [INR]), or standard therapeutic doses of low molecular weight heparin (LMWH), and/or glucocorticoids and immunosuppressants/biologics (e.g., cyclophosphamide, cyclosporine, tacrolimus, rituximab, etc.).
2. Meet all four criteria for catastrophic APS:

i) Involvement of three or more organs, systems, and/or tissues; ii) Development of manifestations within one week; iii) Histopathological confirmation of small vessel occlusion in at least one organ or tissue; iv) Positive antiphospholipid antibodies (aPL).

4. Inflammatory Myopathy (IM)

1. Meet the 2017 EULAR/ACR classification criteria for inflammatory myopathy (including dermatomyositis, polymyositis, anti-synthetase syndrome, and immune-mediated necrotizing myopathy).
2. Have positive myositis-specific autoantibodies.
3. For participants with muscle involvement: a Manual Muscle Test-8 (MMT-8) score <142, and at least two of the following five core abnormalities: Physician Global Assessment ≥2, Patient Global Assessment ≥2, or extramuscular disease activity score ≥2; Health Assessment Questionnaire (HAQ) total score ≥0.25; muscle enzyme levels ≥1.5 times the upper limit of normal; or MMT-8 ≥142 but with active interstitial lung disease (ground-glass opacities on HRCT).

5. Sjögren's Syndrome (SS)

1. Meet the 2016 ACR/EULAR classification criteria for Sjögren's syndrome.
2. Have a EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score ≥5.
3. Have positive anti-SSA/Ro antibodies.
4. Have inadequate response to conventional therapy or disease relapse after remission. Conventional therapy includes glucocorticoids (at full or pulse doses), two or more immunosuppressants, or biologic agents for at least 6 months, including cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, leflunomide, methotrexate, belimumab, telitacicept, and rituximab.

6. Anti-Neutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis (AAV)

1. Meet the 2022 ACR/EULAR classification criteria for ANCA-associated vasculitis (AAV), including microscopic polyangiitis, granulomatosis with polyangiitis, and eosinophilic granulomatosis with polyangiitis.
2. Have a history of or currently positive ANCA.
3. Have a Birmingham Vasculitis Activity Score (BVAS) ≥15 (total score 63).
4. Have inadequate response to conventional therapy or disease relapse after remission. Conventional therapy includes glucocorticoids (at full or pulse doses), two or more immunosuppressants, or biologic agents for at least 6 months, including cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, leflunomide, methotrexate, belimumab, telitacicept, and rituximab.

Exclusion Criteria:

Study participants who meet any of the following criteria will be excluded from the study:

1. Any medical condition that, in the opinion of the investigator, would contraindicate participation in the study, such as a life-threatening illness.
2. Decreased organ function reserve not attributable to the primary disease:

   a) Neutrophil count <1×10⁹/L; lymphocyte count <0.3×10⁹/L; hemoglobin <70 g/L; platelet count <50×10⁹/L; b) Alanine aminotransferase (ALT) >3 × upper limit of normal (ULN); aspartate aminotransferase (AST) >3 × ULN; total bilirubin >2 × ULN; c) Creatinine clearance <40 mL/min; estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m²; or serum creatinine >2.5 mg/dL; d) Left ventricular ejection fraction (LVEF) <45% as measured by echocardiography; e) Oxygen saturation <92% on room air.
3. History of alcohol or substance abuse within the past 24 weeks.
4. History of malignancy other than B-cell lymphoma.
5. Presence of infections including human immunodeficiency virus (HIV), hypogammaglobulinemia, T-cell deficiency, syphilis, chronic hepatitis B or C, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
6. Known active tuberculosis (TB) infection or active bacterial infection.
7. History of myocardial infarction, coronary angioplasty or stenting, unstable angina, clinically significant arrhythmia, or other clinically significant cardiac disease within 6 months prior to screening.
8. Symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to screening, except in cases of antiphospholipid syndrome (APS).
9. History of severe allergic reaction to any component of cellular therapy or other immunotherapeutic agents.
10. Prior organ transplant requiring ongoing immunosuppressive therapy.
11. Concurrent participation in another clinical trial that may interfere with disease assessment or study treatment.
12. Prior treatment with CD19- and/or BCMA-targeted therapy or any CAR-T cell product; except in cases where prior therapy is deemed to have clearly failed (e.g., no response, short duration of response, or disease progression) as assessed by the investigator, the current disease state warrants the study treatment, and there is no clear evidence that toxicity from prior therapy would compromise the safety of the current study.
13. Severe psychiatric disorder or significant cognitive impairment.
14. Pregnancy, lactation, or planned pregnancy.
15. Any other condition that, in the judgment of the investigator, would make the participant unsuitable for enrollment in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities of BCT301 | 28 days
  Adverse events occurring within 28 days post-infusion that were possibly, probably, or definitely related to BCT301 cell injection (per NCI-CTCAE v5.0).

SECONDARY OUTCOMES:
Efficacy of refractory systemic lupus erythematosus（SLE）- The change of SLEDAI-2K | 90, 180, 360 days
  The primary efficacy endpoint will be the change from baseline in the SLEDAI-2K score. The SLEDAI-2K is a validated index for assessing SLE disease activity, with scores ranging from 0 to 105. A higher score indicates worse disease activity.
Efficacy of refractory SLE-The change of PGA | 90, 180, 360 days
  The Physician Global Assessment (PGA) will be used to evaluate overall SLE disease activity. The PGA is a clinician's determination of disease activity based on history and physical exam, independent of laboratory results. It is scored on a scale from 0 to 3, where a higher score indicates worse disease activity.
Efficacy of refractory SLE-The change of SF36 | 90, 180, 360 days
  The SF-36 health survey will be employed as a patient-reported outcome to assess health-related quality of life. This 36-item questionnaire generates scores from 0 to 100 across eight health domains and two summary components (Physical and Mental). A lower score indicates a worse health state
Efficacy of refractory SLE-The change of antibodies | 90, 180, 360 days
  Changes in autoantibody titers (e.g., anti-dsDNA) will be assessed as a serological outcome. A higher autoantibody titer reflects more severe underlying immunologic activity
Efficacy of refractory systemic sclerosis (SSc)-The change of mRSS | 90, 180, 360 days
  The modified Rodnan Skin Score (mRSS) will be the primary endpoint to assess skin disease activity. The mRSS evaluates skin thickness in 17 body areas, with each scored from 0 (normal) to 3 (severe thickening). The total score ranges from 0 to 51, where a higher score indicates worse skin involvement and a poorer prognosis.
Efficacy of refractory SSc-The change of CRISS | 90, 180, 360 days
  The Combined Response Index for Systemic Sclerosis (CRISS) will be used as the primary composite endpoint. This index calculates a probability of improvement (score from 0.0 to 1.0) by integrating changes in skin thickness (mRSS), physician and patient global assessments, functional ability (HAQ-DI), and the absence of new organ damage. A higher score indicates a better treatment response, while a score of 0 indicates treatment failure.
Efficacy of refractory SSc-The change of antibodies | 90, 180, 360 days
  Changes in autoantibody titers (e.g., anti-SCL70) will be assessed as a serological outcome. A higher autoantibody titer reflects more severe underlying immunologic activity.
Efficacy of refractory Antiphospholipid Syndrome (APS)-new onset thrombotic event | 90, 180, 360 days
  The primary efficacy endpoint is the time to first new objectively confirmed arterial or venous thrombotic event. The occurrence of a new thrombotic event is considered a treatment failure, as it directly demonstrates the failure of the therapy.
Efficacy of refractory APS-The change of antibodies | 90, 180, 360 days
  Reduction in titers of antiphospholipid antibodies (aCL, anti-β2GPI, and LA) will be assessed as a key biomarker of response. A decrease in these antibody levels is interpreted as evidence of a positive immunologic treatment effect.
Efficacy of refractory APS-The change of platelet | 90, 180, 360 days
  In patients with baseline thrombocytopenia, an increase in platelet count is considered a positive indicator of treatment efficacy, signifying control of the underlying autoimmune and consumptive processes in APS.
Efficacy of refractory APS- The change of fibrinogen | 90、180、360 days
  In patients with baseline hypofibrinogenemia, an increase in fibrinogen level is considered a positive indicator of treatment efficacy
Efficacy of refractory inflammatory myositis (IM)-The change of TIS | 90, 180, 360 days
  Total Improvement ScoreThe Total Improvement Score (TIS) will be the primary endpoint to define treatment response. The TIS is a composite score (range 0-15) quantifying improvement from baseline across six core domains: muscle strength, physical function, physician and patient global assessments, muscle enzymes, and extramuscular activity. A TIS of ≥ 20 is defined as a clinically meaningful treatment response, with a higher score indicating a greater magnitude of improvement.
Efficacy of refractory IM-The change of CK | 90, 180, 360 days
  Serum Creatine Kinase (CK) level will be assessed as a key biomarker of muscle inflammation. A reduction in CK from baseline, is a defined indicator of positive biochemical treatment response.
Efficacy of refractory IM-The change of antibodies | 90, 180, 360 days
  Reduction in titers of antibodies (e.g. anti-MDA5) will be assessed as a key biomarker of response. A decrease in these antibody levels is interpreted as evidence of a positive immunologic treatment effect.
Efficacy of refractory Sjögren's Disease（SjD）-The change of ESSDAI | 90, 180, 360 days
  The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) will be the primary endpoint to assess systemic disease activity. The ESSDAI scores 12 organ domains, with a total range from 0 (no activity) to 123 (maximal activity). A reduction in the ESSDAI score of ≥3 points from baseline defines a clinically meaningful treatment response, indicating effective suppression of systemic disease.
Efficacy of refractory SjD- Achieving STAR response or not | 90, 180, 360 days
  The Sjögren's Tool for Assessing Response (STAR) will be used as a key patient-reported outcome. The STAR quantifies symptom burden on a scale from 0 (none) to 10 (worst imaginable). A decrease from baseline of ≥1 point in the STAR score defines a clinically meaningful treatment response, indicating a significant reduction in the patient's experience of core symptoms like dryness, fatigue, and pain.
Efficacy of refractory SjD-The change of antibodies | 90, 180, 360 days
  Changes in autoantibody titers (e.g., anti-SSA) will be assessed as a serological outcome. A reduction in titer is considered a favorable immunologic response to therapy.
Efficacy of refractory SjD-The change of immune globulin | 90, 180, 360 days
  Changes in immune globulin will be assessed as a serological outcome. A reduction in titer is considered a favorable immunologic response to therapy.
Efficacy of refractory ANCA associated vasculitis (AAV)-The change of BVAS | 90, 180, 360 days
  The Birmingham Vasculitis Activity Score (BVAS) will be the primary endpoint to assess disease activity. The BVAS quantifies new or worsening vasculitis symptoms across nine organ systems. The total score ranges from 0 (no activity) to over 50, where a higher score indicates worse disease. A reduction in BVAS, particularly to 0, defines treatment response.
Efficacy of refractory AAV-The change of antibody | 90, 180, 360 days
  Serial quantitative ANCA titers (anti-PR3 and anti-MPO) will be assessed as a serological biomarker of response. A significant decrease in ANCA titer is considered a favorable indicator of treatment efficacy.
pharmacokinetic (PK) | 0-28 days
  time to peak (Tmax)
pharmacokinetic (PK) | 0-28 days
  peak concentration (Cmax)
pharmacokinetic (PK) | 0-28 days
  area under the concentration-time curve
pharmacokinetic (PK) | 0-90 days
  area under the concentration-time curve
pharmacodynamic (PD) | 0-28 days
  The count of B cells in peripheral blood post-infusion.

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.